CLINICAL TRIAL: NCT07025122
Title: Fatigue in Multiple Sclerosis and Its Relationship to Inflammatory and Neurodegenerative Markers of the Disease
Acronym: MITOFATIGUE
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital, Martin (Other)
Collaborators: Comenius University (Other)
Responsible Party: Sponsor
Other Study IDs: ID68/2024; VEGA 01/0092/22 (Other Grant/Funding Number: Grant of The Ministry of Education, Research, Development and Youth of the Slovak Republic)
Record Dates: First submitted 2024-11-23; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2024-11

CONDITIONS: Fatigue in Multiple Sclerosis; Multiple Sclerosis; Neurofilaments Light Chains; GFAP; HLA DRB 1501; BCL6 (rs969625); OS9 (rs701006)
Keywords: fatigue, mitochondriopathy, neurofilaments, GFAP, genetics; intergenic variant near BCL6; intronic variant in OS9
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — HLA antigens
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- newly diagnosed multiple sclerosis patients: Newly diagnosed multiple sclerosis patients will be tested before initiation of any immunomodulatory treatment. Tests will be repeated 12 months later.
- All newly diagnosed patients fulfilling McDonal 2017 criteria will be invited to participate.: All newly diagnosed patients fulfilling McDonal 2017 criteria will be invited to participate. Tests will be performed before starting any immunomodulatory treatment. The tests will be performed yearly after initiation of their treatment and evaluated accordingly. Effectivity of the treatment will be evaluated traditionally using NEDA-3 criteria on a yearly base.
  Control group will consist of healthy volunteers. They will be tested ones after entering the study. The tests will include Fatigue questionnaires, sNfL, sGFAP, mitochondrial activity and genetics.

SUMMARY:
The study is focused on several independent quantifiable biomarkers (sNfL, sGFAP, mitochondrial activity, genetics and fatigue tests) to obtain more detailed information about MS and its progression. Based on the results, investigator will further attempt to predict the course of the disease and manage the therapy more effectively to prevent worsening of the patient's condition.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic inflammatory and neurodegenerative disease of the CNS, leading to non-traumatic neurological impairment in young people. Disability progression in MS is commonly recognized as the disability worsening occurring in patients with progressive MS or in the absence of relapse activity in relapsing progressing MS. This process can begin early in the disease and is not always halted by current therapeutics. The ability to accurately select between active, active progressive and nonactive progressive patients is crucial.

The aim of the proposed study is to use a multimodal approach to achieve better diagnosis and more accurate prediction of disease progression in an individual patient. The diagnostic modalities will include the evaluation of fatigue questionnaires (FIS, ESS, HADS, RAND-36), biomarkers examination: serum neurofilament light chain (sNfL) and glial fibrillary acidic protein (sGFAP), and mitochondrial respiratory capacity.

The fatigue questionnaire battery is considered an advanced examination that is not commonly performed in MS patients. The Fatigue Impact Scale (FIS) is a tool used to assess the impact of fatigue on various aspects of a patient's life. This questionnaire measures the extent to which fatigue affects physical, cognitive, and psychosocial functioning and helps quantify the severity of fatigue. The Epworth Sleepiness Scale (ESS) is a simple questionnaire used to measure daytime sleepiness, helping to differentiate increased fatigue in patients from potential sleep disorders. Additionally, HADS and RAND-36 is included in the study to rule out potential associations of fatigue with other external influences.

NfL is known to be an excellent biomarker of focal inflammatory activity but lacks the ability to reflect the pathology that drives disease progression. Neurodegeneration and astrocytic activation can be quantified by glial fibrillary acidic protein (sGFAP). Previous research revealed, that higher levels of sGFAP correlated with subsequent progression, particularly in nonactive patients, whereas sNfL reflected acute disease activity in patients with MS at high risk of underlying progressive pathology.

Mitochondria, traditionally recognized as cellular 'powerhouses' due to their pivotal role in energy production, have emerged as multifunctional organelles at the intersection of bioenergetics, metabolic signalling, and immunity. Investigators propose mitochondria as the leading immune organelles, drawing parallels with the broader immune system in their functions of antigen presentation, immune regulation, and immune response. Investigators also consider mitochondria's ability to detect and release danger signals, regulate immune functions, and engage in intercellular crosstalk. Investigators plan to analyse mitochondrial function by means of high-resolution respirometry with the Oroboros O2k in all study participants.

The human leukocyte antigen (HLA) DRB1*1501, which has been consistently associated with MS nearly in all populations will be evaluated in all participants of the study. The HLA-DRB1*15:01 haplotype is of importance in the interaction between B and T cells in MS patients, while two autosomal genome-wide significant MS risk alleles significantly alter the distribution B-cell subsets. Investigators are planning to test an intergenic variant near BCL6 (rs969625), associated with high MS risk and decreased naive/memory ratios, and an intronic variant in OS9 (rs701006) corresponded to low MS risk.

The study is focused on several independent quantifiable parameters to obtain more detailed information about MS and its progression. Based on the results, investigators will further attempt to predict the course of the disease and manage the therapy more effectively to prevent worsening of the patient's condition.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of multiple sclerosis using McDonald2017 criteria Patients indicated to immunomodulatory treatment

Exclusion Criteria:

Multimorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients newly diagnosed with multiple sclerosis will be invited to participate in observational prospective study before starting any immunomodulatory treatment. The tests will be repeated on yearly base. Results of studied biomarkers will be evaluate and compare with clinical tests results (EDSS, relapse rate and MRI outcome - NEDA-3).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantification of fatigue and comparision with sNfL, sGFAP, and mitochondrial activity | The patients will be tested yearly. All markers will be evaluated prospectively. The Time Frame is from date of randomization up to 5 years
  Baseline:
  * Tests of serum biomarkers (NfL,GFAP), mitochondrial activity using Oroboros, and questionnaires (FIS, ESS, HANDS, RAND)
  * Genetic tests: the HLA-DRB1*15:01 haplotype, an intergenic variant near BCL6 (rs969625) and an intronic variant in OS9 (rs701006)
  * Characteristics of patient´s disease - neurological disability using EDSS, relapses, MRI activity will be recorded
  Follow- up:
  Patients will be evaluated every 6 months, involving standardized neurological examination. Burden of the disease will be evaluated prospectively.
  Number of relapses will be evaluated yearly and annualized relapse rate will be calculated. EDSS score will be evaluated every 6 months. MRI activity will be tested yearly. Levels of NfL" and GFAP, mitochondrial activity, and questionnaires will also be tested yearly.
  Effectiveness of the disease modifying treatment will be evaluated continuously up to 5 years since the onset.

SECONDARY OUTCOMES:
Correlation of genetic characteristics, biomarkers, fatigue tests, and mitochondrial status with the disease burden. | 5 years after the last reqruited patient
  Calculation of NEDA-3 in each clinical year. Correlation of clinical characteristics with NfL, GFAP, mitochondrial functioning, and genetic determinants to evaluate disease burden
  Time Frame Jan/2024 1-12/2025 1-12/2026 Reqruitement of MS patients, collection o biomarkers and results of fatigue tests. EDSS and MRI recorded yearly. Disease modiying treatment according to slovak rules www.nczis.gov
  1-12/2027 1-12/2028 Statistical evaluation, publication of results Statistical evaluation, publication o results

CONTACTS AND LOCATIONS:
Overall Officials: Petra Hnilicová, PhD Ing, Study Chair — Comenius University; Ema Kantorová, prof MD PhD, Principal Investigator — UHMartin and Comenius University; Martin Kolísek, assoc.prof RNDr, Dr.rer.nat., Study Chair — Comenius University; Štefan Sivák, prof.MD, PhD, Study Director — UHMartin and Comenius University; Natália Huňarová, Mgr, doctorand, Study Chair — Comenius University; Andrea Ižarik Verešpejová, Mgr, doctorand, Study Chair — Comenius University; Daniel Čierny, associate prof, MD, PhD, Study Chair — UHMartin and Comenius University; Vladimír Nosáľ, associate prof, MD, PhD, Study Chair — UHMartin, Comenius University
Locations (1):
- University Hospital in Martin, Comenius University, Martin, Slovakia, Slovakia

IPD SHARING:
Plan to Share IPD: Yes
* to inform scientific community about the plant
  * to find cooperators
Supporting Information: Study Protocol
Time Frame: March 2025
Access Criteria: E-mail communication is preferable access

REFERENCES:
- See also: Jessenius Faculty of Medicine in Martin, Comenius University Bratislava — http://www.jfmed.uniba.sk